CLINICAL TRIAL: NCT03106805
Title: Early (4th Week) Versus Late (6thweek) Interval Postpartum Copper Intrauterine Device Insertion: a Randomized Controlled Trial
Brief Title: Early Versus Late Interval Postpartum Copper Intrauterine Device Insertion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAIUD
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Contraception Behavior
Keywords: intrauterine device
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insertion by the end of the 4th week postpartum (Experimental)
  Interventions: Procedure: early insertion
- insertion by the end of the 6th week postpartum (Active Comparator)
  Interventions: Procedure: late insertion

INTERVENTIONS:
Procedure: early insertion — insertion at 4th postpartum week
  Arms: insertion by the end of the 4th week postpartum
Procedure: late insertion — insertion at 6th postpartum week
  Arms: insertion by the end of the 6th week postpartum

SUMMARY:
The optimal interval between pregnancies is debated, but a duration greater than 11-18 months has been suggested as reducing complications in the subsequent pregnancy. Improved birth spacing can be a key benefit use of long-acting reversible contraception, but delay to initiation can still be problematic.So women who have recently given birth can be cost-effectively targeted for family planning education and engagement because often they are already connected with health professionals

ELIGIBILITY:
Inclusion Criteria:

Delivered (vaginal or Cesarean) a singleton living baby ≥28weeks gestation. Women desire birth spacing for one year or more. Women who will accept to participate in the study and follow up.

Exclusion Criteria:

1. Known uterine anomalies.
2. Women with previous ectopic pregnancy.
3. Presence of postpartum pyrexia.
4. Women with history of postpartum hemorrhage in the last delivery either primary or secondary.
5. Retained products of conception.
6. History of previous uterine perforation.
7. Anticipation of difficulty of subsequent follow-up with the women.
8. Women with uncontrolled diabetes and hypertension.
9. Women who wish to use other contraceptive methods.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The number of participants use the device | 6 weeks
  number of women place the intrauterine device within 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shachar BZ, Mayo JA, Lyell DJ, Baer RJ, Jeliffe-Pawlowski LL, Stevenson DK, Shaw GM. Interpregnancy interval after live birth or pregnancy termination and estimated risk of preterm birth: a retrospective cohort study. BJOG. 2016 Nov;123(12):2009-2017. doi: 10.1111/1471-0528.14165. Epub 2016 Jul 13. PMID 27405702